CLINICAL TRIAL: NCT00005079
Title: Timing of Breast Cancer Surgery, Menstrual Cycle and Prognosis
Brief Title: Timing of Menstrual Cycle and Surgery in Treating Premenopausal Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: UCLA-9810046; CDR0000067686 (Registry Identifier: PDQ (Physician Data Query)); UCSD-985772; NCI-G00-1724
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2003-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: conventional surgery

SUMMARY:
RATIONALE: The timing of breast cancer surgery within the menstrual cycle may affect outcome. It is not yet known if treatment is more effective during the initial or final phase of the menstrual cycle.

PURPOSE: Phase III trial to determine the effect of menstrual cycle phase at surgery in treating premenopausal women who have stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if the timing of breast surgery during the menstrual cycle impacts disease recurrence, progression, or death among different racial groups in premenopausal women with stage I, II, or III breast cancer.
* Determine if definitive breast cancer surgeries (e.g., lumpectomy or mastectomy) performed during the follicular phase result in poorer prognosis (recurrence, disease progression, or death) compared with surgeries performed during the midcycle or luteal phases in this patient population.

OUTLINE: This is a multicenter study.

Patients undergo either fine needle aspiration concurrently with definitive breast surgery (mastectomy or lumpectomy) or needle-directed excisional biopsy followed by definitive breast surgery.

Patients undergo serum collection for hormonal analysis preoperatively, 24 hours post operatively, at days 7 and 14, and at 3 months and urine collection for hormonal analysis beginning 24 hours prior to surgery and continuing daily until the onset of the next menses.

Patients complete a 30-minute telephone interview regarding medical, family, occupational, and reproductive history and lifestyle habits (e.g., diet, exercise, or environmental exposures). Beginning 24 hours prior to surgery and continuing until the onset of the next menses, patients complete a menstrual cycle journal indicating the start and length of menses.

Patients undergoing mastectomy are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter. Patients undergoing adjuvant therapy are followed every 3 months for 3 years and then every 6 months thereafter or every 4 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 400 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I, II, or III primary breast cancer undergoing breast surgery

  * Invasive disease (e.g., lobular or ductal)
  * No bilateral disease
* No distant metastases
* Premenopausal

  * Regular menses (no amenorrhea of more than 90 days) without hormone replacement
  * Documented last menstrual period
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Premenopausal

Sex:

* Female

Menopausal status:

* See Disease Characteristics

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior malignancies
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No preoperative chemotherapy

Endocrine therapy:

* No concurrent hormonal replacement therapy
* No concurrent interruptive oral contraceptive use of less than 3 months

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* No prior hysterectomy and/or bilateral oophorectomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena R. Chang, MD, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California